CLINICAL TRIAL: NCT03725904
Title: Daytime Profile of Salivary Progesterone During the Mid-luteal Phase of IVF and FET Cycles
Brief Title: Daytime Profile of Salivary Progesterone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peter Humaidan (Other)
Collaborators: Boston IVF (Other)
Responsible Party: Sponsor-Investigator, Peter Humaidan, Professor, Regionshospitalet Viborg, Skive
Organization: Regionshospitalet Viborg, Skive (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Saliva1
Record Dates: First submitted 2018-10-26; First posted 2018-10-31 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2018-10

CONDITIONS: Infertility, Female
Keywords: Progesterone; Saliva; IVF; Frozen embryo transfer
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IVF/FET (Experimental)
  Interventions: Diagnostic Test: Progesterone analysis in saliva

INTERVENTIONS:
Diagnostic Test: Progesterone analysis in saliva — Analysis of salava progesterone

SUMMARY:
The aim of this study is to perform a 12-hour profile of free saliva progesterone during the luteal phase after fresh and frozen embryo transfer. If progesterone levels in saliva samples show a constant level during daytime, this non-invasive measurement can be used in future ART patients with insufficient progesterone levels who might benefit from additional exogenous progesterone supplementation.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years
* One or two good quality embryos for transfer on day 5.
* BMI >18,5 <30 kg/m²

Exclusion Criteria:

* No good quality embryos for transfer
* Uterine abnormalities
* One ovary
* Oocyte donation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Levels of free progesterone in saliva | 12 hours

SECONDARY OUTCOMES:
Clinical pregnancy rate | 8 weeks
  Ultrasound detected gestational sack divided with number of embryo transfer
Ongoing pregnancy rate | 12 weeks
  Viable pregnancy after gestational week 12+0

CONTACTS AND LOCATIONS:
Locations (1):
- Fertility Clinic Regional Hospital Skive, Skive, Denmark

IPD SHARING:
Plan to Share IPD: No